CLINICAL TRIAL: NCT01589952
Title: Pilot Study of First Line Combination Treatment With Low Dose Pegylated Interferon and Entecavir in Treatment-naïve Patients With Chronic Hepatitis B.
Brief Title: Pegylated Interferon and Entecavir Combination in Chronic Hepatitis B (CHB)
Acronym: Bangabandhu
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Mamun-Al-Mahtab, Associate Professor of Hepatology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BB1
Record Dates: First submitted 2012-05-01; First posted 2012-05-02 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Hepatitis B
Keywords: Pegalyted interferon; Entecavir
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pegylated Interferon, Entecavir (Experimental): 'Pegylated Interferon, Entecavir' arm will consist of 20 chronic hepatitis B patients who will receive Pegylated Interferon 90 micro gms subcutaneously once weekly in combination with entecavir 0.5 mg orally once daily for 24 weeks
  Interventions: Drug: Pegalyted interferon, Entecavir

INTERVENTIONS:
Drug: Pegalyted interferon, Entecavir — Pegalyted interferon: 90 micro gms subcutaneously once weekly for 24 weeks Entecavir: 0.5 mg orally once daily for 24 weeks
  Other Names: Pegasys; Pegin; Optipeg; Baraclude; Enviral; Teviral; Barcavir; Tecavir

SUMMARY:
According to published literature, treatment with pegylated interferon (Peg-IFN) is associated with end of treatment response in treatment naive patients with chronic hepatitis B (CHB). It has antiviral as well as anti-fibrotic properties and treatment with Peg-IFN results in improvement of liver histology and down regulation of progression to cirrhosis of liver. Peg-IFN is administered for a finite duration. The major limitation of Peg-IFN is that only 30-49% patients are benefited by this anti-viral drug. Another potent anti-viral drug, entecavir (ETV), on the other hand, reduces HBV replication in most patients, but causes improvement of liver histology in only 30%, possibly because of its lack of immune modulatory ability like Peg-IFN. Also, ETV treatment is associated with several complications like emergence of HBV mutant. The aim of this study is to assess whether the combination of these two 'unique' anti-viral drugs offer the best possible outcome to treatment-naïve CHB patients, in terms of treatment response (virological and biochemical), treatment cost and duration and adverse events.

DETAILED DESCRIPTION:
Aims & Objectives:

Peg-IFN has five unique features, namely (i) finite duration of administration, (ii) anti-viral effect, (iii) immune-modulation, (iv) anti-fibrotic effect and (v) delayed virologic response off-treatment. However these benefits come at a cost i.e. the drug is expensive and there are several known adverse events.

ETV is a potent nucleoside analogue (Nuc), which has minimal resistance compared to most other Nucs. It is efficient for inducing rapid decline of HBV DNA. However ETV has no known immune modulatory or anti-fibrotic effect and therefore off-treatment response or improvement of hepatic histology is not expected with ETV. Similar to other NUCs, there is no defined duration of administration of ETV.

It has been hypothesized that if lower-dose of Peg-IFN can be given in combination with ETV in treatment-naïve CHB patients, they are likely to benefit most from the 'best of both the drugs' in terms of viral and biochemical responses, treatment cost and duration and adverse events.

The project aims to evaluate the outcome of first-line combination treatment with 'lower-dose Peg-IFN plus ETV' in treatment-naïve CHB patients to see whether this combination may be further evaluated and eventually recommended as first-line management for HBV related chronic liver diseases (CLD).

Research Question:

Although the best treatment option for CHB is not clarified yet, certain therapeutic concepts can be derived from the experience of treating patients with chronic hepatitis C (CHC) and human immunodeficiency virus (HIV) infections. A major advancement in treating CHC and HIV infections has been the development of first-line combination therapy.

The research question of this study is whether the first-line combination treatment with 'lower-dose Peg-IFN plus ETV' is effective and beneficial in treatment-naïve CHB patients and whether this combination may be evaluated further and eventually recommended as the preferred first-line management for HBV related CLD.

Methodology:

Ethical consideration

Ethical approval for the study has been obtained from the Ethical Committee at Bangabandhu Sheikh Mujib Medical University. The study will be performed according to principle of the 'Declaration of Helsinki' of 1975 maintaining all the requisites and norms of 'good clinical practice' (GCP).

This will be a prospective, open label, interventional clinical study. The first 20 (twenty) treatment-naive hepatitis B virus 'e' antigen (HBeAg) positive CHB patients with treatment indication, presenting from July 2011 onwards, who can afford the treatment with Peg-IFN and who voluntarily agree to be part of the study will be recruited. Signed voluntary consent in Bengali will be obtained from each participant.

Patients will receive peg-IFN (90 µgms) sub-cutaneously once weekly for 24 weeks in combination with ETV (0.5 mg) once daily orally for the same duration. Administration of Peg-IFN will be supervised and patients will be evaluated regularly both clinically and with biochemical and haematological parameters for early detection and management of adverse event(s) if any.

Virologic and biochemical parameters will be tested (i) at baseline, (ii) at end of treatment (i.e. at 24 weeks) and (iii) at 12 weeks off-treatment.

These will include HBeAg, HBV DNA and serum alaninetransaminase (ALT). Besides for assessment of liver status, patients will undergo ultrasonography (USG) of hepato-biliary system (HBS), endoscopy of upper gastrointestinal tract (UGIT) and if possible liver biopsy or fibroscan of liver at baseline.

Data analysis All data will be collected using pre-designed questionnaire and preserved in a safe place. Data will be analysed using SPSS programme.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg positive >6 months, HBeAg positive or negative, serum ALT normal or raised and HBV DNA >1000 copies/ml in HBeAg negative or HBV DNA >10000 copies/ml in HBeAg positive.

Exclusion Criteria:

* Coinfection with HCV or HIV, cirrhosis of liver

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-02 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Combination of half dose and reduced duration pegalyted interferon in combination with entecavir achieves biochemical and virologic response in chronic hepatitis B | 6 months
  Combination of half dose and reduced duration pegalyted interferon in combination with entecavir achieves biochemical and virologic response in chronic hepatitis B

CONTACTS AND LOCATIONS:
Overall Officials: Mamun A Mahtab, MSc MD FACG, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh